CLINICAL TRIAL: NCT01789489
Title: Contribution of 3D Sonohysterography and Virtual Hysteroscopy in Exploration of the Uterine Cavity in Comparison to the Diagnostic Hysteroscopy.
Brief Title: 3D Ultrasound - Based Hysteroscopy Versus Virtual Hysteroscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/12
Record Dates: First submitted 2013-01-10; First posted 2013-02-12 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Endometrial or Uterine Pathology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 dimensional sonohysterography (Active Comparator): 3 dimensional sonohysterography
  Interventions: Device: Medison Accuvix V20, sonde 3D5-9EK (Endovaginal 3 dimensional echography)
- Standard hysteroscopy (Active Comparator): Standard hysteroscopy
  Interventions: Device: Medison Accuvix V20, sonde 3D5-9EK (Endovaginal 3 dimensional echography)

INTERVENTIONS:
Device: Medison Accuvix V20, sonde 3D5-9EK (Endovaginal 3 dimensional echography)

SUMMARY:
To prove that the 3 dimensional sonohysterography is, at least, as effective as the diagnostic hysteroscopy in examining the uterine cavity.

ELIGIBILITY:
Inclusion Criteria:

- Diagnostic hysteroscopy prescribed either for a case of infertility or in case of doubt of endometrial / uterine pathology suspected by ultrasound or hysterography.

Exclusion Criteria:

* Current Pregnancy.
* Genital infection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Polyps, fibrosis, atrophy, hypertrophy and other uterine pathology detected by 3D sonohysterography (Accuracy of uterine cavity exploration by 3D sonohysterography) | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie FAY, MD, Study Chair — Hôpital FOCH 40, rue Worth 92150 Suresnes
Locations (1):
- Hôpital FOCH, Suresnes, France